CLINICAL TRIAL: NCT00573794
Title: A Multicenter, Open-Label Study of the Human Anti-TNF Monoclonal Antibody Adalimumab to Evaluate the Long Term Safety and Tolerability of Repeated Administration of Adalimumab in Subjects With Ulcerative Colitis
Brief Title: Long-term Open-label Safety and Efficacy Study of Adalimumab in Subjects With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-223; 2007-004157-28 (EudraCT Number)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab 40 mg EOW/EW (Experimental): Open-label adalimumab 40 mg every other week (EOW) or every week (EW). Participants who entered from an open-label cohort continued their previous dosing regimen of adalimumab EOW or EW; participants who entered from a double-blind cohort received adalimumab EOW.
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — adalimumab prefilled syringes administered as subcutaneous injection EW or EOW
  Other Names: ABT-D2E7; HUMIRA

SUMMARY:
To assess the long-term safety and maintenance of response of adalimumab in subjects with ulcerative colitis who participated in and successfully completed M06-826 (NCT00385736) or M06-827 (NCT00408629).

ELIGIBILITY:
Inclusion Criteria:

* Subject must have successfully enrolled and completed either study M06-826 (NCT00385736) or study M06-827 (NCT00408629)
* Subject is judged to be in generally good health as determined by the principal investigator

Exclusion Criteria:

* Subject has not responded to weekly adalimumab therapy in M06-826 (NCT00385736) or M06-827 (NCT00408629)
* Subject considered by the investigator, for any reason, to be an unsuitable candidate
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2007-11-28 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Background] Colombel JF, Sandborn WJ, Ghosh S, Wolf DC, Panaccione R, Feagan B, Reinisch W, Robinson AM, Lazar A, Kron M, Huang B, Skup M, Thakkar RB. Four-year maintenance treatment with adalimumab in patients with moderately to severely active ulcerative colitis: Data from ULTRA 1, 2, and 3. Am J Gastroenterol. 2014 Nov;109(11):1771-80. doi: 10.1038/ajg.2014.242. Epub 2014 Aug 26. PMID 25155227
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- See also: Related Info. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 592 subjects were randomized and received at least 1 dose of study drug (safety population); 7 subjects enrolled at 3 noncompliant sites were excluded from the analyses (Intent-to-treat 1 [ITT-1] population; N=585).
Period: Overall Study
Arm/Group | Adalimumab 40 mg EOW/EW
Started (ITT-1: All subjects who received ≥1 dose of study drug excluding 7 subjects at noncompliant sites.) | 585
Completed | 255
Not Completed | 330
Not completed — Adverse Event | 81
Not completed — Withdrew Consent | 90
Not completed — Lost to Follow-up | 13
Not completed — Protocol Violation | 6
Not completed — Lack of Efficacy | 94
Not completed — Other | 46

BASELINE CHARACTERISTICS:
Population: ITT-1: All subjects who received ≥1 dose of study drug excluding 7 subjects at noncompliant sites.
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 585
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214
  Male | 371

OUTCOME MEASURES:

1. Primary Outcome: Partial Mayo Score: Change From Baseline Over Time
Description: The Partial Mayo score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Partial Mayo score indicates improvement.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 584
units on a scale
  Baseline | 2.5 (2.02)
  Change from Baseline to Week 48: number analyzed (Participants) | 512
  Change from Baseline to Week 48 | -0.2 (2.04)
  Change from Baseline to Week 96: number analyzed (Participants) | 432
  Change from Baseline to Week 96 | -0.4 (1.78)
  Change from Baseline to Week 144: number analyzed (Participants) | 371
  Change from Baseline to Week 144 | -0.5 (2.06)
  Change from Baseline to Week 192: number analyzed (Participants) | 292
  Change from Baseline to Week 192 | -0.6 (1.84)
  Change from Baseline to Week 240: number analyzed (Participants) | 179
  Change from Baseline to Week 240 | -0.8 (1.79)
  Change from Baseline to Week 292: number analyzed (Participants) | 73
  Change from Baseline to Week 292 | -0.7 (2.05)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | -1.0 (1.97)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | -2.0 (1.00)

2. Primary Outcome: Mayo Score: Change From Baseline Over Time
Description: The Mayo score ranges from 0 (normal or inactive disease) to 12 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding, endoscopy, and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo score indicates improvement.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 583
units on a scale
  Baseline | 3.5 (2.72)
  Change from Baseline to Week 48: number analyzed (Participants) | 493
  Change from Baseline to Week 48 | -0.3 (2.64)
  Change from Baseline to Week 96: number analyzed (Participants) | 422
  Change from Baseline to Week 96 | -0.5 (2.49)
  Change from Baseline to Week 144: number analyzed (Participants) | 360
  Change from Baseline to Week 144 | -0.8 (2.73)
  Change from Baseline to Week 192: number analyzed (Participants) | 277
  Change from Baseline to Week 192 | -0.8 (2.52)
  Change from Baseline to Week 240: number analyzed (Participants) | 168
  Change from Baseline to Week 240 | -1.0 (2.40)
  Change from Baseline to Week 292: number analyzed (Participants) | 72
  Change from Baseline to Week 292 | -0.9 (2.84)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | -1.3 (2.87)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | -2.0 (1.73)

3. Secondary Outcome: Percentage of Participants With Remission Per Partial Mayo Score Over Time
Description: The Partial Mayo score (Mayo score without endoscopy) ranges from 0 (normal or inactive disease) to 9 (severe disease) and is calculated as the sum of 3 subscores (stool frequency, rectal bleeding and physician's global assessment [PGA]), each of which ranges from 0 (normal) to 3 (severe disease). Remission was defined as Partial Mayo score ≤ 2 with no subscore > 1.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with evaluable data at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 585
percentage of participants
  Baseline: number analyzed (Participants) | 584
  Baseline | 52.4
  Week 48: number analyzed (Participants) | 513
  Week 48 | 61.2
  Week 96: number analyzed (Participants) | 433
  Week 96 | 69.3
  Week 144: number analyzed (Participants) | 372
  Week 144 | 75.0
  Week 192: number analyzed (Participants) | 293
  Week 192 | 74.7
  Week 240: number analyzed (Participants) | 180
  Week 240 | 77.2
  Week 292: number analyzed (Participants) | 73
  Week 292 | 76.7
  Week 340: number analyzed (Participants) | 23
  Week 340 | 73.9
  Week 388: number analyzed (Participants) | 3
  Week 388 | 100

4. Secondary Outcome: Mayo Endoscopy Subscore: Change From Baseline Over Time
Description: The Mayo Endoscopy subscore ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo Endoscopy subscore indicates improvement.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 583
units on a scale
  Baseline | 1.1 (0.94)
  Change from Baseline to Week 48: number analyzed (Participants) | 493
  Change from Baseline to Week 48 | -0.1 (0.95)
  Change from Baseline to Week 96: number analyzed (Participants) | 422
  Change from Baseline to Week 96 | -0.1 (1.02)
  Change from Baseline to Week 144: number analyzed (Participants) | 360
  Change from Baseline to Week 144 | -0.2 (0.93)
  Change from Baseline to Week 192: number analyzed (Participants) | 277
  Change from Baseline to Week 192 | -0.3 (0.98)
  Change from Baseline to Week 240: number analyzed (Participants) | 168
  Change from Baseline to Week 240 | -0.3 (0.97)
  Change from Baseline to Week 292: number analyzed (Participants) | 72
  Change from Baseline to Week 292 | -0.3 (1.03)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | -0.3 (1.18)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | 0.0 (1.00)

5. Secondary Outcome: Mayo Rectal Bleeding Subscore: Change From Baseline Over Time
Description: The Mayo Rectal Bleeding subscore ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo Rectal Bleeding subscore indicates improvement.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 584
units on a scale
  Baseline | 0.4 (0.68)
  Change from Baseline to Week 48: number analyzed (Participants) | 512
  Change from Baseline to Week 48 | -0.1 (0.73)
  Change from Baseline to Week 96: number analyzed (Participants) | 432
  Change from Baseline to Week 96 | -0.0 (0.63)
  Change from Baseline to Week 144: number analyzed (Participants) | 371
  Change from Baseline to Week 144 | -0.1 (0.74)
  Change from Baseline to Week 192: number analyzed (Participants) | 292
  Change from Baseline to Week 192 | -0.1 (0.69)
  Change from Baseline to Week 240: number analyzed (Participants) | 179
  Change from Baseline to Week 240 | -0.2 (0.63)
  Change from Baseline to Week 292: number analyzed (Participants) | 73
  Change from Baseline to Week 292 | -0.2 (0.76)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | -0.2 (0.80)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | -1.0 (1.00)

6. Secondary Outcome: Mayo Physician's Global Assessment of Disease Severity Subscore: Change From Baseline Over Time
Description: The Mayo Physician's Global Assessment of Disease Severity subscore ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo Physician's Global Assessment of Disease Severity subscore indicates improvement.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 584
units on a scale
  Baseline | 0.8 (0.81)
  Change from Baseline to Week 48: number analyzed (Participants) | 512
  Change from Baseline to Week 48 | -0.1 (0.89)
  Change from Baseline to Week 96: number analyzed (Participants) | 432
  Change from Baseline to Week 96 | -0.2 (0.84)
  Change from Baseline to Week 144: number analyzed (Participants) | 371
  Change from Baseline to Week 144 | -0.2 (0.89)
  Change from Baseline to Week 192: number analyzed (Participants) | 292
  Change from Baseline to Week 192 | -0.2 (0.82)
  Change from Baseline to Week 240: number analyzed (Participants) | 179
  Change from Baseline to Week 240 | -0.3 (0.82)
  Change from Baseline to Week 292: number analyzed (Participants) | 73
  Change from Baseline to Week 292 | -0.2 (0.79)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | -0.3 (0.88)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | -0.7 (0.58)

7. Secondary Outcome: Mayo Stool Frequency Subscore: Change From Baseline Over Time
Description: The Mayo Stool Frequency subscore ranges from 0 (normal) to 3 (severe disease). A negative change in Mayo Stool Frequency subscore indicates improvement.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 584
units on a scale
  Baseline | 1.3 (1.01)
  Change from Baseline to Week 48: number analyzed (Participants) | 512
  Change from Baseline to Week 48 | -0.1 (0.89)
  Change from Baseline to Week 96: number analyzed (Participants) | 432
  Change from Baseline to Week 96 | -0.2 (0.84)
  Change from Baseline to Week 144: number analyzed (Participants) | 371
  Change from Baseline to Week 144 | -0.2 (0.89)
  Change from Baseline to Week 192: number analyzed (Participants) | 292
  Change from Baseline to Week 192 | -0.2 (0.82)
  Change from Baseline to Week 240: number analyzed (Participants) | 179
  Change from Baseline to Week 240 | -0.3 (0.86)
  Change from Baseline to Week 292: number analyzed (Participants) | 73
  Change from Baseline to Week 292 | -0.3 (1.00)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | -0.5 (0.99)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | -0.3 (0.58)

8. Secondary Outcome: Inflammatory Bowel Disease Questionnaire (IBDQ): Change From Baseline Over Time
Description: The IBDQ is a 32-item questionnaire that assesses how the subject felt during the 2 weeks before the measurement time point. Questions are related to symptoms the subject might have had as a result of UC, how the subject felt in general, how the subject's mood was, and social and work problems the subject might have that resulted from UC. An increase in IBDQ score indicates less impact of UC on the subject's life. The responses to each question range from 1 (significant impairment) to 7 (no impairment), with the total score ranging from 32 (very poor) to 224 (perfect health-related quality of life).
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 572
units on a scale
  Baseline | 176.0 (34.45)
  Change from Baseline to Week 48: number analyzed (Participants) | 485
  Change from Baseline to Week 48 | 2.1 (28.91)
  Change from Baseline to Week 96: number analyzed (Participants) | 412
  Change from Baseline to Week 96 | 4.7 (28.73)
  Change from Baseline to Week 144: number analyzed (Participants) | 355
  Change from Baseline to Week 144 | 5.2 (30.64)
  Change from Baseline to Week 192: number analyzed (Participants) | 279
  Change from Baseline to Week 192 | 7.6 (28.66)
  Change from Baseline to Week 240: number analyzed (Participants) | 174
  Change from Baseline to Week 240 | 11.2 (25.98)
  Change from Baseline to Week 292: number analyzed (Participants) | 70
  Change from Baseline to Week 292 | 14.8 (27.36)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | 14.6 (28.12)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | 11.0 (12.53)

9. Secondary Outcome: 36-Item Short Form Health Survey Version 2 (SF-36) Mental Component Score: Change From Baseline Over Time
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (mental [MCS] and physical [PCS]). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 (poorest health) to 100 (best health) scale with higher scores indicating better health status or functioning.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 575
units on a scale
  Baseline | 47.1 (10.16)
  Change from Baseline to Week 48: number analyzed (Participants) | 498
  Change from Baseline to Week 48 | -0.7 (9.61)
  Change from Baseline to Week 96: number analyzed (Participants) | 423
  Change from Baseline to Week 96 | 0.3 (9.64)
  Change from Baseline to Week 144: number analyzed (Participants) | 360
  Change from Baseline to Week 144 | 0.0 (9.52)
  Change from Baseline to Week 192: number analyzed (Participants) | 286
  Change from Baseline to Week 192 | 0.1 (9.41)
  Change from Baseline to Week 240: number analyzed (Participants) | 178
  Change from Baseline to Week 240 | 0.7 (7.86)
  Change from Baseline to Week 292: number analyzed (Participants) | 71
  Change from Baseline to Week 292 | 1.8 (8.13)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | 1.8 (6.81)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | -7.3 (5.58)

10. Secondary Outcome: 36-Item Short Form Health Survey Version 2 (SF-36) Physical Component Score: Change From Baseline Over Time
Description: as for outcome 9
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 575
units on a scale
  Baseline | 49.3 (8.06)
  Change from Baseline to Week 48: number analyzed (Participants) | 498
  Change from Baseline to Week 48 | 0.7 (6.98)
  Change from Baseline to Week 96: number analyzed (Participants) | 423
  Change from Baseline to Week 96 | 1.2 (6.26)
  Change from Baseline to Week 144: number analyzed (Participants) | 360
  Change from Baseline to Week 144 | 1.1 (7.08)
  Change from Baseline to Week 192: number analyzed (Participants) | 286
  Change from Baseline to Week 192 | 1.3 (7.46)
  Change from Baseline to Week 240: number analyzed (Participants) | 178
  Change from Baseline to Week 240 | 2.2 (6.23)
  Change from Baseline to Week 292: number analyzed (Participants) | 71
  Change from Baseline to Week 292 | 2.5 (7.03)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | 3.0 (8.71)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | 8.4 (2.00)

11. Secondary Outcome: Work Productivity and Activity Impairment: General Health Version 2.0 (WPAI:GH) Work Time Missed Because of Ulcerative Colitis: Change From Baseline Over Time
Description: The WPAI:GH questionnaire was used to assess work and activity impairment due to symptoms of ulcerative colitis in the last 7 days. The self-administered questionnaire measures the effect of the subject's health problems on work and daily activities in the previous week, specifically, the number of hours missed from work due to health problems, how much the subject's health problems affected work productivity, and how much the subject's health problems affected regular activities. Low scores indicate little or no impact of health problems on work and activities, and a negative change in the WPAI score indicates improvement.
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: percent of work time missed
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 375
percent of work time missed
  Baseline | 4.5 (15.42)
  Change from Baseline to Week 48: number analyzed (Participants) | 294
  Change from Baseline to Week 48 | 1.6 (24.04)
  Change from Baseline to Week 96: number analyzed (Participants) | 245
  Change from Baseline to Week 96 | -0.2 (18.41)
  Change from Baseline to Week 144: number analyzed (Participants) | 213
  Change from Baseline to Week 144 | 0.9 (20.19)
  Change from Baseline to Week 192: number analyzed (Participants) | 170
  Change from Baseline to Week 192 | 0.2 (19.05)
  Change from Baseline to Week 240: number analyzed (Participants) | 109
  Change from Baseline to Week 240 | -1.1 (17.21)
  Change from Baseline to Week 292: number analyzed (Participants) | 47
  Change from Baseline to Week 292 | 8.2 (30.65)
  Change from Baseline to Week 340: number analyzed (Participants) | 16
  Change from Baseline to Week 340 | 6.4 (24.96)
  Change from Baseline to Week 388: number analyzed (Participants) | 2
  Change from Baseline to Week 388 | 0.0 (0.00)

12. Secondary Outcome: WPAI:GH Impairment While Working: Change From Baseline Over Time
Description: as for outcome 11
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: percent of work time impaired
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 388
percent of work time impaired
  Baseline | 16.7 (20.73)
  Change from Baseline to Week 48: number analyzed (Participants) | 315
  Change from Baseline to Week 48 | 1.1 (22.45)
  Change from Baseline to Week 96: number analyzed (Participants) | 262
  Change from Baseline to Week 96 | -1.9 (20.86)
  Change from Baseline to Week 144: number analyzed (Participants) | 233
  Change from Baseline to Week 144 | -0.2 (24.11)
  Change from Baseline to Week 192: number analyzed (Participants) | 177
  Change from Baseline to Week 192 | -2.9 (24.04)
  Change from Baseline to Week 240: number analyzed (Participants) | 119
  Change from Baseline to Week 240 | -4.0 (21.40)
  Change from Baseline to Week 292: number analyzed (Participants) | 52
  Change from Baseline to Week 292 | -3.8 (25.45)
  Change from Baseline to Week 340: number analyzed (Participants) | 16
  Change from Baseline to Week 340 | -13.8 (26.04)
  Change from Baseline to Week 388: number analyzed (Participants) | 2
  Change from Baseline to Week 388 | -15.0 (21.21)

13. Secondary Outcome: WPAI:GH Overall Work Impairment: Change From Baseline Over Time
Description: as for outcome 11
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: percent of overall work impairment
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 373
percent of overall work impairment
  Baseline | 20.1 (24.30)
  Change from Baseline to Week 48: number analyzed (Participants) | 294
  Change from Baseline to Week 48 | 1.2 (28.15)
  Change from Baseline to Week 96: number analyzed (Participants) | 244
  Change from Baseline to Week 96 | -2.7 (24.99)
  Change from Baseline to Week 144: number analyzed (Participants) | 212
  Change from Baseline to Week 144 | -0.8 (28.05)
  Change from Baseline to Week 192: number analyzed (Participants) | 168
  Change from Baseline to Week 192 | -2.6 (26.69)
  Change from Baseline to Week 240: number analyzed (Participants) | 109
  Change from Baseline to Week 240 | -5.0 (24.1)
  Change from Baseline to Week 292: number analyzed (Participants) | 47
  Change from Baseline to Week 292 | 1.4 (35.53)
  Change from Baseline to Week 340: number analyzed (Participants) | 16
  Change from Baseline to Week 340 | -7.3 (12.05)
  Change from Baseline to Week 388: number analyzed (Participants) | 2
  Change from Baseline to Week 388 | -15.0 (21.21)

14. Secondary Outcome: WPAI:GH Activity Impairment: Change From Baseline Over Time
Description: as for outcome 11
Time Frame: Baseline (Week 0), Weeks 48, 96, 144, 192, 240, 292, 340, 388
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: percent activity impaired
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 550
percent activity impaired
  Baseline | 21.4 (24.00)
  Change from Baseline to Week 48: number analyzed (Participants) | 479
  Change from Baseline to Week 48 | 1.1 (24.14)
  Change from Baseline to Week 96: number analyzed (Participants) | 405
  Change from Baseline to Week 96 | -1.6 (21.80)
  Change from Baseline to Week 144: number analyzed (Participants) | 351
  Change from Baseline to Week 144 | -0.7 (23.65)
  Change from Baseline to Week 192: number analyzed (Participants) | 267
  Change from Baseline to Week 192 | -2.1 (20.91)
  Change from Baseline to Week 240: number analyzed (Participants) | 171
  Change from Baseline to Week 240 | -3.4 (18.63)
  Change from Baseline to Week 292: number analyzed (Participants) | 68
  Change from Baseline to Week 292 | -1.5 (19.79)
  Change from Baseline to Week 340: number analyzed (Participants) | 23
  Change from Baseline to Week 340 | -9.6 (11.86)
  Change from Baseline to Week 388: number analyzed (Participants) | 3
  Change from Baseline to Week 388 | -16.7 (15.28)

15. Secondary Outcome: Colectomy Rate
Description: The colectomy rates were estimated using Kaplan-Meier methodology based on the time to first colectomy.
Time Frame: 5 years
Population: ITT-1 population
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 585
percentage of participants | 3.88

16. Secondary Outcome: Health Care Resource Utilization (HCRU): Cumulative Number of Unscheduled Utilizations
Description: The HCRU assesses the frequency of unscheduled outpatient visits, emergency room visits, or hospitalizations due to ulcerative colitis since the last visit. The cumulative number of unscheduled utilizations over the course of the study is presented.
Time Frame: 5 years
Population: ITT-1 population
Measure: Number; unit: cumulative number of utilizations
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 585
cumulative number of utilizations
  Physician | 561
  Emergency Room | 43
  Hospital Admission | 65
  Days in Hospital | 435

17. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Time Frame: From first dose of study drug until 70 days after the last dose of study drug (up to 398 weeks)
Population: Safety analysis set: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 592
Participants
  Any TEAE | 496
  Any TESAE | 158

18. Secondary Outcome: Hematology: Mean Change From Baseline to Final Values in Hemoglobin
Description: Blood samples for laboratory tests were performed at each study visit after questionnaires and vital sign determinations.
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in the safety analysis set with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 575
g/L | -0.1 (16.02)

19. Secondary Outcome: Hematology: Mean Change From Baseline to Final Values in Hematocrit
Description: as for outcome 18
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in the safety analysis set with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 575
Percentage of red blood cells | 0.013 (0.0472)

20. Secondary Outcome: Hematology: Mean Change From Baseline to Final Values in Red Blood Cell Count, Platelet Count, White Blood Cell Count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils
Description: as for outcome 18
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in the safety analysis set with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: cells * 10^9/L
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 575
cells * 10^9/L
  Red blood cell count | 0.03 (0.416)
  Platelet count: number analyzed (Participants) | 572
  Platelet count | -10.5 (96.98)
  White blood cell count | 0.41 (2.704)
  Neutrophils: number analyzed (Participants) | 572
  Neutrophils | 0.164 (2.4225)
  Lymphocytes: number analyzed (Participants) | 572
  Lymphocytes | 0.155 (0.8270)
  Monocytes: number analyzed (Participants) | 572
  Monocytes | 0.051 (0.2203)
  Eosinophils: number analyzed (Participants) | 572
  Eosinophils | 0.002 (0.1602)
  Basophils: number analyzed (Participants) | 572
  Basophils | 0.009 (0.0586)

21. Secondary Outcome: Clinical Chemistry: Mean Change From Baseline to Final Values in Alanine Aminotransferase, Aspartate Aminotransferase, and Alkaline Phosphatase
Description: as for outcome 18
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in the safety analysis set with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 581
U/L
  Alanine aminotransferase: number analyzed (Participants) | 579
  Alanine aminotransferase | 3.7 (22.03)
  Aspartate aminotransferase: number analyzed (Participants) | 579
  Aspartate aminotransferase | 2.6 (28.13)
  Alkaline phosphatase | -0.2 (34.65)

22. Secondary Outcome: Clinical Chemistry: Mean Change From Baseline to Final Values in Total Bilirubin, Creatinine, and Uric Acid
Description: as for outcome 18
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in ITT-1 population with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 581
μmol/L
  Total bilirubin | -1.0 (5.35)
  Creatinine | 2.4 (13.18)
  Uric acid | 7.6 (65.52)

23. Secondary Outcome: Clinical Chemistry: Mean Change From Baseline to Final Values in Blood Urea Nitrogen, Inorganic Phosphate, Calcium, Sodium, Potassium, Glucose, Cholesterol, and Triglycerides
Description: as for outcome 18
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in the safety analysis set with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 581
mmol/L
  Blood urea nitrogen | 0.32 (1.409)
  Inorganic phosphate | -0.003 (0.2312)
  Calcium | -0.012 (0.1185)
  Sodium | -0.0 (2.49)
  Potassium | 0.07 (0.424)
  Glucose | 0.05 (1.334)
  Cholesterol | -0.025 (0.8853)
  Triglycerides | 0.178 (1.2800)

24. Secondary Outcome: Clinical Chemistry: Mean Change From Baseline to Final Values in Albumin and Total Protein
Description: as for outcome 18
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in the safety analysis set with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 581
g/L
  Albumin | -0.4 (3.85)
  Total protein | 0.7 (18.99)

25. Secondary Outcome: Clinical Chemistry: Mean Change From Baseline to Final Values in High-sensitivity C-reactive Protein
Description: as for outcome 18
Time Frame: Baseline (Week 0), final value (up to 5 years)
Population: Participants in the safety analysis set with both Baseline and visit values.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Adalimumab 40 mg EOW/EW
Number analyzed (Participants) | 575
mg/L | 0.382 (15.1489)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 398 weeks).
Description: TEAEs and TESAEs are defined as any adverse event or serious adverse event with onset or worsening from the time that the first dose of adalimumab is administered until 5 half-lives (70 days) have elapsed following discontinuation of adalimumab administration. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Adalimumab 40 mg EOW/EW
Serious Adverse Events (participants affected / at risk) | 158/592
Other Adverse Events (participants affected / at risk) | 391/592
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg EOW/EW (N=592)
ANAEMIA (Blood and lymphatic system disorders) | 6
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY MEDIASTINAL (Blood and lymphatic system disorders) | 1
AORTIC VALVE STENOSIS (Cardiac disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 2
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1
TACHYCARDIA (Cardiac disorders) | 1
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 1
ADRENAL HAEMORRHAGE (Endocrine disorders) | 1
GOITRE (Endocrine disorders) | 1
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
ANAL FISTULA (Gastrointestinal disorders) | 1
COLITIS (Gastrointestinal disorders) | 3
COLITIS ULCERATIVE (Gastrointestinal disorders) | 34
COLON DYSPLASIA (Gastrointestinal disorders) | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 1
GASTROINTESTINAL DYSPLASIA (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1
PSEUDOPOLYPOSIS (Gastrointestinal disorders) | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2
RECTAL PERFORATION (Gastrointestinal disorders) | 1
RECTAL POLYP (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 1
DRUG INTOLERANCE (General disorders) | 1
DYSPLASIA (General disorders) | 1
MULTIMORBIDITY (General disorders) | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1
POLYP (General disorders) | 1
PYREXIA (General disorders) | 1
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 2
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1
PORTAL HYPERTENSION (Hepatobiliary disorders) | 1
ABDOMINAL ABSCESS (Infections and infestations) | 2
ABSCESS OF SALIVARY GLAND (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 3
APPENDICITIS (Infections and infestations) | 5
APPENDICITIS PERFORATED (Infections and infestations) | 1
CHRONIC SINUSITIS (Infections and infestations) | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1
COLONIC ABSCESS (Infections and infestations) | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1
DIARRHOEA INFECTIOUS (Infections and infestations) | 1
DIVERTICULITIS (Infections and infestations) | 1
HERPES ZOSTER (Infections and infestations) | 2
HERPES ZOSTER MENINGITIS (Infections and infestations) | 1
INFECTION (Infections and infestations) | 2
INJECTION SITE ABSCESS (Infections and infestations) | 1
INJECTION SITE CELLULITIS (Infections and infestations) | 1
LUNG ABSCESS (Infections and infestations) | 1
ORCHITIS (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 2
PNEUMONIA (Infections and infestations) | 11
PNEUMONIA BACTERIAL (Infections and infestations) | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 1
PYELONEPHRITIS (Infections and infestations) | 2
PYELONEPHRITIS ACUTE (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2
URINARY TRACT INFECTION (Infections and infestations) | 1
ANIMAL BITE (Injury, poisoning and procedural complications) | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 1
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1
FALSE POSITIVE TUBERCULOSIS TEST (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 1
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 3
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 5
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
SYMPATHETIC POSTERIOR CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 1
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CERVIX CARCINOMA STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
GALLBLADDER ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1
DEMYELINATION (Nervous system disorders) | 1
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 1
NERVE COMPRESSION (Nervous system disorders) | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 2
BIPOLAR I DISORDER (Psychiatric disorders) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
PSYCHOTIC BEHAVIOUR (Psychiatric disorders) | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 1
DYSURIA (Renal and urinary disorders) | 1
URETEROLITHIASIS (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
MENORRHAGIA (Reproductive system and breast disorders) | 2
OVARIAN CYST (Reproductive system and breast disorders) | 1
PROSTATISM (Reproductive system and breast disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
UTERINE CYST (Reproductive system and breast disorders) | 1
ALLERGIC RESPIRATORY SYMPTOM (Respiratory, thoracic and mediastinal disorders) | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1
NASAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 2
HENOCH-SCHONLEIN PURPURA (Skin and subcutaneous tissue disorders) | 1
ABORTION INDUCED (Surgical and medical procedures) | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
HAEMORRHAGIC INFARCTION (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg EOW/EW (N=592)
ABDOMINAL PAIN (Gastrointestinal disorders) | 38
COLITIS ULCERATIVE (Gastrointestinal disorders) | 180
DIARRHOEA (Gastrointestinal disorders) | 46
NAUSEA (Gastrointestinal disorders) | 34
FATIGUE (General disorders) | 35
BRONCHITIS (Infections and infestations) | 40
INFLUENZA (Infections and infestations) | 42
SINUSITIS (Infections and infestations) | 53
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 58
URINARY TRACT INFECTION (Infections and infestations) | 31
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 115
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 62
BACK PAIN (Musculoskeletal and connective tissue disorders) | 40
HEADACHE (Nervous system disorders) | 46
COUGH (Respiratory, thoracic and mediastinal disorders) | 41
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 33
RASH (Skin and subcutaneous tissue disorders) | 42
HYPERTENSION (Vascular disorders) | 37

LIMITATIONS AND CAVEATS:
Efficacy data after Week 292 should be interpreted with caution because less than 10% of subjects were under observation beyond Week 292.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.